CLINICAL TRIAL: NCT02099422
Title: The Randomized TOPIC Study : Timing of Optimal Platelet Inhibition After Acute Coronary Syndrome
Brief Title: Timing of Optimal Platelet Inhibition After Acute Coronary Syndrome
Acronym: TOPIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital de la Timone (Other)
Responsible Party: Principal Investigator, CUISSET Thomas, MD-PHD, Hôpital de la Timone
Other Study IDs: APHM-011; 2013-A01168-37 (Other: AFSSAPS)
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Acute Coronary Syndrome; Coronary Stenting; Antiplatelet Therapy
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of two antiplatelet strategies between months 1 and 12 after coronary stenting for ACS. Efficiency and tolerance évaluation

ELIGIBILITY:
Inclusion Criteria:

* ACS and coronary stenting one month ago

Exclusion Criteria:

* age under 18 and pregnancy

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ACS treated by coronary stent implantation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
combined ischemic and hemorragic endpoint | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Timone hospital . Sc CARDIOLOGIE. Rue saint Pierre., Marseille, France